CLINICAL TRIAL: NCT07273344
Title: A Systems Immunology Approach to Characterize the Immune Response in Sepsis and Its Long-term Complications
Brief Title: A Study on How the Immune System Responds to Sepsis and Its Long-term Effects
Acronym: HEAL-SEPSIS
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Research Council (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL010169
Record Dates: First submitted 2025-11-14; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Sepsis
Keywords: observational; sepsis; cohort study; immune endotypes; endotypes; immunotypes; post-sepsis syndrome
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Whole blood, plasma, peripheral blood mononuclear cells (PBMC's), PAXgene tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — This study involves no interventions beyond scheduled blood collection.

SUMMARY:
Sepsis occurs when an infection, caused by bacteria, a virus, or a fungus, enters the body and throws the immune system out of balance. Instead of protecting the body, the immune response may become too strong and start damaging healthy organs, or it may become too weak and fail to control the infection. Both situations can be life-threatening. Even people who survive sepsis may experience long-term health problems, such as new infections, heart and blood vessel diseases, or early death.

This study aims to better understand how the immune system behaves during and after sepsis. We believe that there are different types of immune responses in sepsis, called immunotypes. We will identify these immunotypes by examining substances in the blood and changes in immune cells. We will then study which immunotypes help protect patients and which may cause short- or long-term harm.

Understanding these immunotypes may make it possible in the future to quickly determine what type of immune response a patient with sepsis has. This could help doctors choose the best treatment for each individual patient.

A total of 400 patients with sepsis from the intensive care unit will take part in this study. We will collect blood samples at several time points and gather information about their health. Participants will be followed from their intensive care admission until one year after they return home.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ failure syndrome caused by a dysregulated host response to infection. Despite advances in antimicrobial therapy and intensive care, mortality remains high due to our inability to rebalance the host immune response. Current immunotherapy strategies fail to account for the highly heterogeneous immunopathological mechanisms underlying sepsis. Some patients experience hyperinflammation, others immune paralysis, with these states often coexisting or shifting over time. Moreover, different immunological mechanisms may drive each of these broad patterns of immune dysregulation. Defining patient immunotypes and identifying associated biomarkers is therefore essential for developing targeted immunotherapies. Additionally, the long-term morbidity and mortality following sepsis, potentially driven by lasting epigenetic changes, are poorly understood. A deeper understanding of immunotypes and their impact on both acute and long-term outcomes is essential to improve patient stratification and guide future precision medicine approaches in sepsis.

This study aims to characterize sepsis immunotypes linked to short- and long-term outcomes and identify novel biomarkers and therapeutic targets. This is a multicenter, prospective, observational cohort study. We aim to recruit a cohort of 400 intensive care or medium care patients diagnosed with sepsis, as defined by the Sepsis-3 criteria. No randomization will be performed. Blood samples and clinical data will be collected on the following timepoints: day 0 (within 48 hours of ICU/MC admission), day 3 (±1 day, defined as 3 days after day 0), at hospital discharge (±2 days), and at 3 and 12 months post-discharge (each ±2 weeks). Patients will be retrospectively classified into subgroups according to infection site, as defined by the International Sepsis Forum Consensus Conference definitions. This study involves no interventions beyond scheduled blood collection. The amount of blood drawn at each timepoint will not exceed 40 ml. To minimize additional venipunctures during admission, blood collection will be incorporated into routine clinical care whenever possible. Clinical data at 3 and 12 months post-discharge will be gathered through questionnaires or phone interviews. The only additional travel required for the study is for post-discharge blood collection, which participants can choose to complete at an external Radboudumc-affiliated blood collection site closest to their home. Therefore, for all patients-including those who may be incapacitated during the acute phase of sepsis-the risks and burden associated with participation are considered minimal. Patients will not receive any direct benefit from participating in this study. However, the knowledge gained is expected to guide future sepsis diagnoses, treatment and prediction of health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18years).
* Sepsis 3 criteria: defined as having a suspected or documented infection accompanied by organ dysfunction, represented by a total Sequential Organ Failure Assessment (SOFA-2) score 2 or more for new admissions or as 2 or more point-increase of the total SOFA-2 score for hospitalized patients.

Exclusion Criteria:

* Known chemotherapy-induced or long-term neutropenia.
* Known CD4 counts <400 cells/µL.
* History of primary immunodeficiency
* Chronic intake of corticosteroids (defined as total daily dose equal or greater than 0.4 mg/kg of equivalent prednisone for more than the last 15 days).
* Current use of biologics.
* Solid organ transplant recipients.
* Recipients of allogeneic bone marrow transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU or medium care patients diagnosed with sepsis, as defined by the Sepsis-3 criteria, from the Radboudumc, Canisius Wilhelmina Ziekenhuis, Rijnstate Ziekenhuis, and Jeroen Bosch Ziekenhuis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Classification of hospitalized sepsis patients into distinct immunotypes. | Day 0 (within 48 hours of intensive care unit admission or start of sepsis)
Classification of hospitalized sepsis patients into distinct immunotypes. | Day 3 (defined as 3 days after day 0)
Classification of hospitalized sepsis patients into distinct immunotypes. | At hospital discharge.

SECONDARY OUTCOMES:
Detection of persistent immunotypes at following hospital discharge. | Three months after hospital discharge.
Detection of persistent immunotypes at following hospital discharge. | Twelve months after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai G. Netea, Prof. dr., Study Director — Radboud University Medical Center; Wouter A. van der Heijden, dr., Principal Investigator — Radboud University Medical Center; Peter Pickkers, Prof. dr., Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The HEAL-SEPSIS project will share all pseudonymized IPD used in analyses and publications under restricted access, in accordance with participant consent and intellectual property protections. Privacy and confidentiality obligations prevent unrestricted sharing of full IPD datasets